CLINICAL TRIAL: NCT03230500
Title: Patient Satisfaction and Early Implant Failure of Computer-guided Versus Free- Hand Immediate Implant Placement in Fresh Extraction Sockets in Esthetic Zone, a Randomized Clinical Trial.
Brief Title: Computer Guided Versus Free Hand Immediate Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Safaa Kamel Hussein, Assisstant Lecturer- Prosthodontic Department- Faculty of Dentistry- Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Faculty of Dentistry
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Dental Implants
Keywords: computer guided; immediate implant; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the trial only the outcome assessor will be masked from the intervention or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer guided immediate implant placement (Experimental): For the test group, the computer aided surgical guide will be used for implant drilling and placement.
  Interventions: Procedure: Computer guided implant placement
- Free hand immediate implant placement (Active Comparator): For the control group, free hand implant drilling and placement will be performed guided by the extraction socket walls.
  Interventions: Procedure: Computer guided implant placement

INTERVENTIONS:
Procedure: Computer guided implant placement — Implant will be placed immediately using computer aided surgical guide

SUMMARY:
Patients with remaining root or fractured teeth indicated for extraction in the esthetic zone will be recruited to the study. After extraction of the tooth implant will be placed immediately, implants will be placed either by free hand or computer guided technique. patient satisfaction will be evaluated as primary outcome and early implant failure was evaluated as secondary outcome.

DETAILED DESCRIPTION:
General operative procedures:

Eligible patients will be randomized, at the surgical phase in two groups, study group (in which computer guided implant placement was done using computer aided surgical guide) and comparative group (in which free hand implant placement was done).

Patients of both groups will be subjected to:

Careful clinical examination and medical and dental history taking. CBCT scan will be performed while patients biting on cotton roll to separate the teeth of interest from opposing dentition, moreover cotton rolls will be placed in vestibule for separation of lip and check from teeth of interest.After examination of the CBCT scan, maxillary and mandibular alginate impression will be made for eligible patients.For temporary crown fabrication after the surgery, the tooth or root to be extracted will be modified on the study cast and an artificial tooth will be placed. After that a 2mm hard vacuum sheet will be pressed on the study cast. For the test group (computer guided group), three dimensional (3d) virtual planning of the surgical guide and implant position will be made with the aid of Blue Sky ® implant planning software . After proper selection of implant size, diameter and position, the virtual surgical guide will be exported as a STL file for 3D printing. Before the surgery, adaptation of the surgical guide will be checked on the study cast and a metallic sleeve will be attached at proposed implant position using adhesive.

Intraoperative procedure:

3 days before the surgery, a prophylactic antibiotic will be given to the patient. On the day of surgery, local anaesthesia will be injected and a traumatic extraction of the remaining root or tooth will be performed. For a traumatic extraction, gentle application of a periotome mesio-distally along with slight rotational movement. After extraction, intact labial and palatal socket walls will be checked using periodontal probe for immediate implant placement. For the test group, the computer aided surgical guide will be checked for adaptability and any interference will be removed. After that implant drilling and placement will be performed using the surgical guide. For the control group, free hand implant drilling and placement will be performed guided by the extraction socket walls. For both groups implant primary stability will be checked by application of 35 Ncm2 force using torque wrench After that, the final abutment will be screwed in its position and the temporary crown will be made using the vacuum stent, where a chair side tooth coloured autopolymerizing resin will be injected into the vacuum stent at the proposed implant site. Finally, occlusion will be checked for any functional contact in maximum intercuspation and lateral movement. Any contact with the opposing should be removed and the patient will be instructed to avoid eating or incising on the temporary crown for at least two weeks. Seven days later patients will be recalled for inspection and taking postoperative photos, six months thereafter, the patient will receive a definitive crown.

ELIGIBILITY:
Inclusion Criteria:

Patients with teeth or remaining roots in the esthetic zone and indicated for extraction and replacement with immediate implant.

Sufficient labial bone to avoid labial plate fracture during extraction (at least 1.5-2 mm). This will be confirmed by cone beam computer tomography (CBCT) scan.

Sufficient mesio distal length between the neighbouring natural teeth (at least 7 mm), this will be confirmed on the study cast.

Presence of adjacent teeth to the tooth or remaining root to be extracted.

Exclusion Criteria:

Heavy smokers (more than 2 packs / day). Patients with parafunctional habits (e.g. clenching or bruxism, etc.) Presence of acute infection in the tooth or the remaining root that will be extracted.

Severe overeruption of the opposing teeth to avoid premature contact with the temporary crown during the healing period.

Patients with poor oral hygiene Pregnant women Any systemic condition that may interfere with implant placement and its osseointegration (as uncontrolled diabetes, chemotherapy, radiotherapy. Osteonecrosis…)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 0-6 months
  Patient satisfaction will be assessed through a questionnaire and each question of the questionnaire will be scored by the patients on 10 cm visual analogue scales (VAS)

SECONDARY OUTCOMES:
Early implant failure | 0-6 months
  Early implant failure will be clinically diagnosed by implant loss from mouth which will be detected by visual inspection. Early implant failure will be assessed in the interval between implant placement until functional loading (0-6 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Safaa hussein, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schropp L, Isidor F, Kostopoulos L, Wenzel A. Patient experience of, and satisfaction with, delayed-immediate vs. delayed single-tooth implant placement. Clin Oral Implants Res. 2004 Aug;15(4):498-503. doi: 10.1111/j.1600-0501.2004.01033.x. PMID 15248886
- [Background] Misch CE, Perel ML, Wang HL, Sammartino G, Galindo-Moreno P, Trisi P, Steigmann M, Rebaudi A, Palti A, Pikos MA, Schwartz-Arad D, Choukroun J, Gutierrez-Perez JL, Marenzi G, Valavanis DK. Implant success, survival, and failure: the International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference. Implant Dent. 2008 Mar;17(1):5-15. doi: 10.1097/ID.0b013e3181676059. PMID 18332753
- [Result] Sabir M, Alam MN. Survival of Implants in Immediate Extraction Sockets of Anterior Teeth: Early Clinical Results. J Clin Diagn Res. 2015 Jun;9(6):ZC58-61. doi: 10.7860/JCDR/2015/13631.6123. Epub 2015 Jun 1. PMID 26266220